CLINICAL TRIAL: NCT07172516
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Azetukalner in Depressive Episodes Associated With Bipolar I or II Disorder (Bipolar Depression)
Brief Title: A Randomized Study of Azetukalner Versus Placebo in Depressive Episodes Associated With Bipolar I or II Disorder (Bipolar Depression)
Acronym: X-CEED
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-010-B301
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder
Keywords: Bipolar; XEN1101; Azetukalner
MeSH Terms: conditions — Bipolar Disorder | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azetukalner (Experimental): Azetukalner 20 mg
  Interventions: Drug: Azetukalner
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azetukalner — Azetukalner 20 mg taken orally once a day with food (with the evening meal when possible) for 6 weeks
  Other Names: XEN1101
  Arms: Azetukalner
Drug: Placebo — Placebo taken orally once a day with food (with the evening meal when possible) for 6 weeks
  Arms: Placebo

SUMMARY:
X-CEED is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of azetukalner in adult participants diagnosed with bipolar I or II disorder who are currently in a depressive episode (bipolar depression).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥18 and ≤74 years of age who experienced their first major depressive episode (MDE) prior to 50 years of age.
* Body Mass Index (BMI) ≥18 kg/m2 and ≤40 kg/m2.
* Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR) criteria for bipolar I or II disorder and is currently in a MDE, confirmed using the Mini International Neuropsychiatric Interview (MINI).
* Current MDE must has a duration of ≥4 weeks and ≤12 months.

Key Exclusion Criteria:

* Participant has any type of major depressive disorder (MDD) diagnosis, including MDD with psychotic features, MDD with catatonia, MDD with seasonal pattern, or postpartum depression.
* Participant has any nonbipolar psychiatric diagnosis.
* Participant has a substance use disorder (excluding tobacco) within the 6 months prior to screening visit.
* Participant has a symptomatic eating disorder within the 12 months prior to screening visit.
* Participant has a Young Mania Rating Scale (YMRS) score >12 points at screening visit or randomization.
* Participant has been hospitalized for mania within the 30 days prior to screening visit.
* Participant is considered treatment-resistant in the current bipolar depressive episode, defined as having treatment resistance (no remission) to ≥2 different medications approved by the regional regulatory authority at an adequate dose (per regulatory approved label) and for an adequate duration (at least 6 weeks).
* Participant has had an active suicidal plan/intent within the 6 months prior to screening, presence of suicidal behavior in the last 12 months.
* Participant has self-injurious behavior without intent to die in the 12 months prior to screening.
* Participant has used antidepressants, mood stabilizers, anticonvulsants, antipsychotics, or other prohibited medications within the 1 week or within a period less than 5 times the drug's half-life, whichever is longer prior to randomization.
* Participants with medical conditions that may interfere with the purpose or conduct of the study.
* Participant is pregnant, breastfeeding, or planning to become pregnant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score at Week 6. | Baseline to Week 6

SECONDARY OUTCOMES:
Change from baseline in the Clinical Global Impression of Severity (CGI-S) score at Week 6. | Baseline to Week 6
Change from baseline in the MADRS total score at Week 1. | Baseline to Week 1
Change from baseline in the Snaith-Hamilton Pleasure Scale (SHAPS) total score at Week 6. | Baseline to Week 6

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Noble Clinical Research, Tucson, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Clinical Innovations Inc, Bellflower, California
  - ProScience Research Group, Culver City, California
  - ATP Clinical Research, Orange, California
  - NRC Research Institute, Orange, California
  - Clinical Innovations Inc, Riverside, California
  - PharmaSouth Research, LLC, Coral Gables, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Synexus Clinical Research, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, Decatur, Georgia
  - Denali Health Atlanta, LLC, Stone Mountain, Georgia
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Lumina Clinical Research Center, Cherry Hill, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Neurobehavioral Research Inc, Cedarhurst, New York
  - DelRicht Research, Charlotte, North Carolina
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Elevate Synapsis, LLC, Atascocita, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Eastside Therapeutics Resources, INC dba Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No